CLINICAL TRIAL: NCT02392299
Title: Frailty, Cardiovascular Function and Risk of Falling in Patients Receiving Haemodialysis Treatment
Brief Title: Risk of Falling in Chronic Kidney Disease 5
Status: Completed | Type: Observational
Sponsor: Queen Margaret University (Other)
Collaborators: British Renal Society (Other); British Kidney Patient Association (Unknown)
Responsible Party: Principal Investigator, P KOUFAKI, Research Fellow, Queen Margaret University
Other Study IDs: BUR(14/17)
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Stage 5 Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to explore the relative importance of the frailty and cardiovascular function as potential exercise-modifiable risk factors for falling in patients receiving haemodialysis.

DETAILED DESCRIPTION:
Falls and fall-related injuries in elderly people are common worldwide, and ageing populations will further raise the burden and costs. Within the UK, falls have become a major government target, as they have been responsible for increased injuries and hospital admissions in elderly people.

The fall rate amongst patients on haemodialysis (HD) is much greater than in the general population. There are many well established risk factors for falling, many of which are commonly present in patients on HD, including severe loss of muscle mass, high levels of inactivity, co-existing medical conditions and a high number of medications.

Nonetheless, the main cause of health complications and death in Chronic Kidney Disease (CKD) is due to cardiovascular disease. Cardiovascular disease may result in suboptimal regulation of blood pressure and heart rate during exercise, dialysis therapy, body transfers, and general activities of daily living. Associated symptoms such as dizziness, generalised fatigue, and muscular weakness, are commonly reported and may further predispose patients on HD to balance deficits and falls.

Despite the evidence of high falls rates in patients on HD and the growing number of elderly patients, falls and their associated risk factors have received little research attention.

The aim of this study therefore is explore the relative importance of selected exercise-modifiable risk factors for falling amongst patients on HD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Able to write/speak fluent English
* Stable dialysis

Exclusion Criteria:

* Unstable dialysis and medication treatment
* Lower limb amputees without prothesis
* Unstable cardiac condition
* Suspected or known aneurysm
* Clinically severe left ventricular outflow obstruction
* Critical mitral stenosis
* Critical proximal coronary artery stenosis
* Critical cerebrovascular stenosis
* Pregnancy
* Severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 5 Chronic Kidney Disease patients
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-09; Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Falls incidence | One year

SECONDARY OUTCOMES:
Frailty components | baseline
  muscle strength, balance, gait speed, body composition

OTHER OUTCOMES:
Cardiovascular Function | baseline
  blood pressure, baroreceptor reflexes

CONTACTS AND LOCATIONS:
Overall Officials: Tobia Zanotto, MSc, Principal Investigator — Queen Margaret University
Locations (2):
- United Kingdom (2):
  - Monklands Renal Unit, Airdrie
  - Renal Unit, Falkirk

REFERENCES:
- [Derived] Zanotto T, Mercer TH, van der Linden ML, Rush R, Traynor JP, Petrie CJ, Doyle A, Chalmers K, Allan N, Shilliday I, Koufaki P. The relative importance of frailty, physical and cardiovascular function as exercise-modifiable predictors of falls in haemodialysis patients: a prospective cohort study. BMC Nephrol. 2020 Mar 14;21(1):99. doi: 10.1186/s12882-020-01759-z. PMID 32169050